CLINICAL TRIAL: NCT00958204
Title: Light and Ion Treatment to Enhance Medication Efficacy in Depression
Brief Title: Light, Ion, and Fluoxetine Efficacy (LIFE) in Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H09-01015
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depression; rating scales; RCT; combination treatment; light therapy; negative ion therapy; fluoxetine; antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Light treatment using a fluorescent light box (30 minutes daily) plus a placebo pill every day
  Interventions: Procedure: Light treatment; Drug: Placebo
- 2 (Experimental): Negative ion generator (30 minutes daily) plus 20 mg of fluoxetine per day
  Interventions: Procedure: Negative ion therapy; Drug: Fluoxetine
- 3 (Active Comparator): Light treatment using a fluorescent light box (30 minutes daily) plus 20 mg of fluoxetine per day
  Interventions: Procedure: Light treatment; Drug: Fluoxetine
- 4 (Placebo Comparator): Negative ion generator (30 minutes daily) plus placebo pill every day
  Interventions: Procedure: Negative ion therapy; Drug: Placebo

INTERVENTIONS:
Procedure: Light treatment — Light therapy: from a 10,000 lux fluorescent white light box, for 30 minutes per day upon waking in the morning, for 8 weeks.
  Arms: 1; 3
Procedure: Negative ion therapy — Negative ion therapy: from a negative ion generator with an output of 200 trillion ions per second per cubic centimeter, for 30 minutes per day upon waking in the morning, for 8 weeks
  Arms: 2; 4
Drug: Placebo — Placebo Pill: one oral tablet each day, for 8 weeks.
  Arms: 1; 4
Drug: Fluoxetine — Fluoxetine: 20 mg oral tablet each day, for 8 weeks
  Arms: 2; 3

SUMMARY:
This study will investigate the additional benefits of light and ion therapy as added treatments to an antidepressant (fluoxetine) in subjects with major depressive disorder (MDD), versus treatment with fluoxetine alone. Outcomes will include depressive symptom rating scales and measures of quality of life, work absence and productivity, and use of health care services. The primary hypotheses are that, in patients with nonseasonal major depressive disorder (MDD) of at least moderate severity: 1) bright light therapy or negative ion therapy will be superior to a placebo condition in reducing symptoms of depression, and 2) the combination of fluoxetine and either bright light or negative ion therapy is more effective than either monotherapy condition.

DETAILED DESCRIPTION:
Rationale

Many effective treatments exist for depression, including psychotherapies and antidepressant medications. However, antidepressants are not always effective, and they can produce significant side effects and pose a risk of overdose. Medication can also be expensive, thereby limiting accessibility. Furthermore, many people with MDD prefer to use non-pharmacological treatments. Some studies have found that combination antidepressant and psychotherapy is more effective than either monotherapy in people with chronic forms of MDD. However, evidence-based psychotherapies such as cognitive-behavioural therapy are not widely available within the Canadian health care system.

For these reasons, there is great interest in finding alternative treatments to antidepressants and psychotherapy. Bright light therapy, which is well established as an effective treatment for seasonal affective disorder (SAD), has many attributes that make it highly attractive to use for nonseasonal MDD: it is a safe, well-tolerated, inexpensive, easy to use, non-pharmacological treatment that can be used as monotherapy or combined with medications without the worry of drug-drug interactions. The "gold standard" method for applying light therapy is via a 10,000 lux white fluorescent light box for 30 minutes a day, usually in the early morning upon arising from bed. The mechanism of action of light therapy is still unknown, but major hypotheses involve resynchronizing circadian rhythms and/or restoring neurotransmitter dysfunction. Bright light has predictable phase-shifting effects on circadian rhythms in humans, but studies of light therapy have not consistently demonstrated correlations of phase shift with antidepressant response. Although most of these studies have been done in patients with SAD, there is considerable evidence that nonseasonal MDD is also associated with disturbances in circadian rhythms. Other studies have shown that rapidly depleting serotonin and catecholamines can reverse the antidepressant effects of light therapy in SAD, thereby demonstrating monoaminergic effects of bright light similar to those seen with antidepressants. These chronobiologic and monoaminergic effects of bright light provide a rationale for the use of light therapy in nonseasonal MDD. As well, initial studies have shown that negative ion generators may be an effective treatment for neurovegetative symptoms of SAD, specifically oversleeping, overeating, and fatigability. However, relatively few studies have been conducted of light and ion therapy in nonseasonal MDD. Several systematic reviews of light and ion therapy for nonseasonal MDD have shown some support for efficacy, but these are based on a limited number of small-sample, poorly controlled RCTs.

Research Method

This study is an 8-week, multi-centre, double-blind (subject and rater), randomized, parallel-design trial to assess the efficacy of light and ion therapy when combined with fluoxetine in the treatment of subjects with MDD, compared to treatment with fluoxetine alone. A total of 216 depressed patients meeting entry criteria will be enrolled over a three-year period.

Eligible patients will be randomized to one of four treatment conditions for the entire treatment period (8 weeks):

1. light treatment using a fluorescent light box (30 minutes daily) plus a placebo pill every day; or
2. negative ion generator (30 minutes daily) plus 20 mg of fluoxetine per day; or
3. negative ion generator (30 minutes daily) plus placebo pill every day; or
4. light treatment using a fluorescent light box (30 minutes daily) plus 20 mg of fluoxetine per day.

Half of all devices (light boxes and negative ions) will be deactivated to test placebo conditions.

Outcomes (HAM-D) will be primarily assessed over the telephone by raters blind to treatment assignment. Other outcome measures will be assessed by patient-rated questionnaires administered over the Internet using a secure web site, and by ratings from the treating physician (CGI and Health Economics Assessment).

Statistical Analysis All randomized subjects who have at least one follow-up visit will be included in the analysis based on intent-to-treat. Ineligible subjects who are inappropriately randomized will be excluded from the analysis. Missing data will be imputed using last observation carried forward (LOCF). For the analyses the treatment variables will remain coded and the analysts and investigators will remain blinded to variable identity during analysis and interpretation.

The pre-specified primary efficacy endpoint is the adjusted mean change from baseline to endpoint (8 weeks) in the HAM-D score using LOCF. All comparisons will be analyzed using ANCOVA adjusting for baseline value and centre. The secondary outcomes will also be analyzed using a similar analysis, when appropriate. Post-hoc analyses will also examine observed case data. Categorical data (such as proportions of the sample with adverse events) will be analyzed using chi-square tests or Fisher's test where cell sizes warrant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 19-60 years.
* Patients will meet DSM-IV criteria for major depressive disorder as determined by the mood disorders section of the Mini International Neuropsychiatric Interview (MINI, Sheehan et al, 1998).
* A score of 20 or greater on the Hamilton Depression Rating Scale (Ham-D), indicating at least moderately severe depression.
* Competency to give informed consent.

Exclusion Criteria:

* Pregnant women, lactating women and sexually active women of childbearing potential who are not using medically accepted means of contraception.
* Serious suicidal risks as judged by the clinician and the MINI.
* The following DSM-IV diagnoses (to ensure a homogeneous diagnostic group): organic mental disorders; substance abuse/dependence, including alcohol, active within the last year; schizophrenia, paranoid, or delusional disorders; other psychotic disorders; panic disorder or generalized anxiety disorder, if a primary diagnosis; obsessive-compulsive disorder or post-traumatic stress disorder; bipolar disorder; bulimia nervosa or anorexia nervosa.
* Serious illness including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic and hematologic disease that is not stabilized, or a past history of convulsions.
* Any retinal disease or systemic illness with active retinal involvement (e.g. diabetes) that precludes the use of bright light.
* Patients who have a history of severe allergies and multiple drug adverse reactions.
* Regular or current use of other psychotropic drugs, including lithium and tryptophan.
* Patients treated with beta blocking drugs.
* Hypertensive patients being treated with guanethidine, reserpine, clonidine or methyldopa (because of possible mood-altering effects of those drugs).
* Use of monoamine oxidase inhibitors within 14 days of Visit 1 (to ensure no drug interactions between fluoxetine and MAOIs), or use of heterocyclic antidepressants within 7 days of Visit 1 (to ensure adequate washout period of two weeks between stopping previous drug and start of treatment at Visit 2).
* Previous use of fluoxetine or light therapy.
* Treatment resistance in the current episode, as defined by failure (lack of clinically significant response) of two or more antidepressants given at therapeutic doses for at least 6 weeks.
* Patients who start formal psychotherapy (e.g. cognitive-behavioural or interpersonal psychotherapy) within 3 months of Visit 1, or who plan to initiate such psychotherapy during this study.
* Patients involved in any other form of treatment for depression.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2009-10; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in adjusted HAM-D scores at 2-month follow-up. | 2 months

SECONDARY OUTCOMES:
At 2-month follow-up: clinical response and remission rates, absenteeism and work productivity, adverse events, quality of life, and health services. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Serge Beaulieu, Dr., Study Director — McGill University; Amy HY Cheung, Dr., Study Director — University of Toronto; Alexander J. Kiss, Dr., Study Director — Sunnybrook Health Sciences Centre; Robert D. Levitan, Dr., Study Director — University of Toronto; Anthony J. Levitt, Dr., Study Director — University of Toronto; Erin E. Michalak, Dr., Study Director — University of British Columbia; Rachel L. Morehouse, Dr., Study Director — Dalhousie University; Sagar V. Parikh, Dr., Study Director — University of Toronto; Rajamannar Ramasubbu, Dr., Study Director — University of Calgary; Glenda MacQueen, Dr., Study Director — University of Calgary; Raymond W. Lam, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- UBC Hospital Mood Disorders Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Levitan RD, Levitt AJ, Michalak EE, Morehouse R, Ramasubbu R, Yatham LN, Tam EM, Lam RW. Appetitive Symptoms Differentially Predict Treatment Response to Fluoxetine, Light, and Placebo in Nonseasonal Major Depression. J Clin Psychiatry. 2018 Jul 24;79(4):17m11856. doi: 10.4088/JCP.17m11856. PMID 30063303
- [Derived] Lam RW, Levitt AJ, Levitan RD, Michalak EE, Cheung AH, Morehouse R, Ramasubbu R, Yatham LN, Tam EM. Efficacy of Bright Light Treatment, Fluoxetine, and the Combination in Patients With Nonseasonal Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jan;73(1):56-63. doi: 10.1001/jamapsychiatry.2015.2235. PMID 26580307